CLINICAL TRIAL: NCT01401153
Title: Cross-over Trial Determining the Short-term Effects of Lunch on Children's Cognitive Functioning
Brief Title: Cognition Intervention Study Dortmund
Acronym: CogniDO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Institute of Child Nutrition, Dortmund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: COG0611DO; 03MT110527328495 (Other Grant/Funding Number: Uniscientia Stiftung)
Record Dates: First submitted 2011-07-19; First posted 2011-07-25 (Estimated); Results first posted 2012-11-09 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-10

CONDITIONS: Cognition - Other

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Having lunch/skipping lunch (Experimental): Lunch ad libitum on test day 1 and no lunch on test day 2. Water available on both days.
  Interventions: Other: Skipping lunch
- Skipping lunch/having lunch (Experimental): No lunch on test day 1 and lunch ad libitum on test day 2. Water available on both days.
  Interventions: Other: Skipping lunch

INTERVENTIONS:
Other: Skipping lunch — Just water.

SUMMARY:
Major aim of this study is to add scientifically proven insights into cognitive effects of meals to the existing recommendations for school meals in Germany. As a first step the short-term effects of skipping lunch on children's cognitive functioning in the afternoon will be examined in a cross-over trial. The study is conducted in a large comprehensive school in Gelsenkirchen (Germany) including about 150 children.

DETAILED DESCRIPTION:
Because of cerebral particularities, children may react sensitive to short-term variations of nutrient supply. Therefore, an optimised composition of meals at nutritionally favourable mealtime should be considered for optimal cognitive performance. The increasing implementation of all-day schools in Germany requires the children's catering at school. However, also the number of 'meal skippers' is increasing among children. Thus, the effect of skipping of the midday meal at school on cognitive functioning is examined in this experimental cross-over trial.

As prior intake of food can have an influence on the physiological effect of test meal, the children's dietary intake in the morning is standardized. The intervention is integrated in the usual everyday school life:

9.15 a.m. standardized snack within the frame of the regular break, 9.45 a.m. to 12.25 p.m. everyday school life, 12.25 p.m. either lunch (control) or only a non-caloric beverage (intervention of 'skipping meal'), 12.45 p.m. to 1.15 p.m. regular lunch break, 1.15 p.m. computerized tests of cognitive functioning, 2 p.m. lunch for the 'skipping meal'-group.

Parameters of cognition with relevance to everyday school life are measured by a computerized test battery of the 'Wiener Testsystem'. Usual eating behaviour, sleep behaviour, physical activity, parental education and migration background are determined as control variables by questionnaires for children, parents and teachers. Beside the Body Mass Index, the individual IQ is measured by a paper-pencil-test.

ELIGIBILITY:
Inclusion Criteria:

* All sixth grade students of Gesamtschule Berger Feld with the consent of parents and child

Exclusion Criteria:

* Metabolic diseases or special diet

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2011-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde Kersting, Prof. Dr., Study Director — Research Institute of Child Nutrition, Dortmund

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from a secondary all-day school in Gelsenkirchen, Germany in May 2011
Pre-assignment Details: 161 participants were assessed for eligibility; 40 children refused to participate; thus 121 children started the study; one-week wash out;
Groups:
- Having Lunch: Lunch ad libitum (pasta Bolognese, apple and water)
- Skipping Lunch: No lunch (water)
Period: First Test Day
Arm/Group | Having Lunch | Skipping Lunch
Started | 66 | 55
Completed | 65 | 45
Not Completed | 1 | 10
Not completed — Learning disabilities; illness | 1 | 10
Period: Second Test Day
Arm/Group | Having Lunch | Skipping Lunch
Started | 45 | 65
Completed | 45 | 60
Not Completed | 0 | 5
Not completed — illness | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Having Lunch | Skipping Lunch | Total
Number analyzed (Participants) | 66 | 55 | 121
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 66 | 55 | 121
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 12.7 (0.6) | 12.7 (0.6) | 12.7 (0.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 32 | 64
  Male | 34 | 23 | 57
Region of Enrollment [Number; unit: participants]
  Germany | 66 | 55 | 121

OUTCOME MEASURES:

1. Primary Outcome: Tonic Alertness (Mean Reaction Time)
Description: Mean reaction time to response to a simple visual stimulus without a preceding warning signal
Time Frame: Participants were tested twice with one week wash out (1h after having/skipping lunch)
Population: Complete case analysis
Measure: Median (Inter-Quartile Range); unit: Milliseconds
Groups:
- Having Lunch: Lunch ad libitum
Arm/Group | Having Lunch | Skipping Lunch
Number analyzed (Participants) | 105 | 105
Milliseconds | 281 [254 to 305] | 279 [256 to 308]
Statistical Analysis 1: Comparison: Having Lunch vs Skipping Lunch; Power calculation had been performed; Test type: Non-Inferiority or Equivalence — Power calculation based on parallel group design --> revealed that 68 children are needed to detect a difference of 45ms in the mean reaction time between the groups, with α=.05 and a power of 0.8; p = 0.79, Wilcoxon (Mann-Whitney); Individual differences of both test days compared on group level (having lunch/skipping lunch vs. skipping lunch/having lunch)

2. Primary Outcome: Tonic Alertness (Deviation of Reaction Time)
Description: Deviation of reaction time --> logarithmic standard deviation of the reaction times
Time Frame: Participants were tested twice with one week wash out (1h after having/skipping lunch)
Population: Complete case analysis
Measure: Median (Inter-Quartile Range); unit: Unitless
Arm/Group | Having Lunch | Skipping Lunch
Number analyzed (Participants) | 105 | 105
Unitless | 77 [56 to 101] | 84 [60 to 113]
Statistical Analysis 1: Comparison: Having Lunch vs Skipping Lunch; Test type: Non-Inferiority or Equivalence — No power calculation had been performed based on this measure; p = 0.07, Wilcoxon (Mann-Whitney); [statistical method as in outcome 1, analysis 1]

3. Primary Outcome: Tonic Alertness (Commission Errors)
Description: Reactions when no stimulus had been presented
Time Frame: Participants were tested twice with one week wash out (1h after having/skipping lunch)
Population: Complete case analysis
Measure: Median (Inter-Quartile Range); unit: Commission errors
Arm/Group | Having Lunch | Skipping Lunch
Number analyzed (Participants) | 105 | 105
Commission errors | 2 [0 to 3] | 2 [1 to 4]
Statistical Analysis 1: Comparison: Having Lunch vs Skipping Lunch; Test type: Non-Inferiority or Equivalence — No power calculation had been performed based on this measure; p = 0.61, Wilcoxon (Mann-Whitney); [statistical method as in outcome 1, analysis 1]

4. Primary Outcome: Tonic Alertness (Omission Errors)
Description: Stimuli to which no reaction follows within 1.5s
Time Frame: Participants were tested twice with one week wash out (1h after having/skipping lunch)
Population: Complete case analysis
Measure: Median (Inter-Quartile Range); unit: Omission errors
Arm/Group | Having Lunch | Skipping Lunch
Number analyzed (Participants) | 105 | 105
Omission errors | 0 [0 to 0] | 0 [0 to 1]
Statistical Analysis 1: Comparison: Having Lunch vs Skipping Lunch; Test type: Non-Inferiority or Equivalence — No power calculation had been perfomed based on this measure; p = 0.03, Wilcoxon (Mann-Whitney); [statistical method as in outcome 1, analysis 1]

5. Primary Outcome: Immediate Block Span
Description: Longest sequence correctly reproduced in at least two of three items (the test is a task of reproducing prescribed sequences from two to eight blocks)
Time Frame: Participants were tested twice with one week wash out (1h after having/skipping lunch)
Population: Complete case analysis
Measure: Median (Inter-Quartile Range); unit: Longest sequence correctly reproduced
Groups:
- Skipping Lunch: No lunch (water) o
Arm/Group | Having Lunch | Skipping Lunch
Number analyzed (Participants) | 105 | 105
Longest sequence correctly reproduced | 5 [4 to 5] | 5 [4 to 5]
Statistical Analysis 1: Comparison: Having Lunch vs Skipping Lunch; Test type: Non-Inferiority or Equivalence — No power calculation had been performed based on this measure; p = 0.25, Generalized linear models; The fixed statement considered treatment, test day and the interaction between treatment and test day

6. Primary Outcome: Incorrect Immediate Block Span
Description: Number of sequences incorrectly reproduced
Time Frame: Participants were tested twice with one week wash out (1h after having/skipping lunch)
Population: Complete case analysis
Measure: Median (Inter-Quartile Range); unit: Sequences incorrectly reproduced
Arm/Group | Having Lunch | Skipping Lunch
Number analyzed (Participants) | 105 | 105
Sequences incorrectly reproduced | 2 [1 to 3] | 2 [1 to 3]
Statistical Analysis 1: Comparison: Having Lunch vs Skipping Lunch; Test type: Non-Inferiority or Equivalence — No power calculation had been performed based on this measure; p = 0.70, Generalized linear models

7. Primary Outcome: Correct Immediate Block Span
Description: Number of sequences correctly reproduced
Time Frame: Participants were tested twice with one week wash out (1h after having/skipping lunch)
Population: Complete case analysis
Measure: Median (Inter-Quartile Range); unit: Sequences correctly reproduced
Arm/Group | Having Lunch | Skipping Lunch
Number analyzed (Participants) | 105 | 105
Sequences correctly reproduced | 10 [8 to 12] | 10 [8 to 12]
Statistical Analysis 1: Comparison: Having Lunch vs Skipping Lunch; Test type: Non-Inferiority or Equivalence — No power calculation had been performed based on this measure; p = 0.33, Generalized linear models

8. Primary Outcome: Sequencing Errors
Description: Sequences including all the blocks of a prescribed sequence, but in the wrong order
Time Frame: Participants were tested twice with one week wash out (1h after having/skipping lunch)
Population: Complete case analysis
Measure: Median (Inter-Quartile Range); unit: Sequences with wrong order
Arm/Group | Having Lunch | Skipping Lunch
Number analyzed (Participants) | 105 | 105
Sequences with wrong order | 2 [1 to 3] | 2 [1 to 3]
Statistical Analysis 1: Comparison: Having Lunch vs Skipping Lunch; Test type: Non-Inferiority or Equivalence — No power calculation had been performed based on this measure; p = 0.63, Generalized linear models

9. Primary Outcome: Reactions
Description: Number of total reactions (Subjects have to decide whether a displayed figure is identical with one of four figures shown or not)
Time Frame: Participants were tested twice with one week wash out (1h after having/skipping lunch)
Population: Complete case analysis
Measure: Median (Inter-Quartile Range); unit: Total reactions
Arm/Group | Having Lunch | Skipping Lunch
Number analyzed (Participants) | 105 | 105
Total reactions | 628 [561 to 704] | 638 [574 to 739]
Statistical Analysis 1: Comparison: Having Lunch vs Skipping Lunch; Test type: Non-Inferiority or Equivalence — No power calculation had been performed based on this measure; p = 0.62, Wilcoxon (Mann-Whitney); [statistical method as in outcome 1, analysis 1]

10. Primary Outcome: Percentage Incorrect Reactions
Description: Percentage of incorrect reactions
Time Frame: Participants were tested twice with one week wash out (1h after having/skipping lunch)
Population: Complete case analysis
Measure: Median (Inter-Quartile Range); unit: Incorrect reactions %
Arm/Group | Having Lunch | Skipping Lunch
Number analyzed (Participants) | 105 | 105
Incorrect reactions % | 4.7 [2.6 to 7.7] | 5.3 [3.4 to 9.3]
Statistical Analysis 1: Comparison: Having Lunch vs Skipping Lunch; Test type: Non-Inferiority or Equivalence — No power calculation had been performed based on this measure; p = 0.11, Wilcoxon (Mann-Whitney); [statistical method as in outcome 1, analysis 1]

11. Primary Outcome: Number Correct Reactions
Description: Number of correct reactions
Time Frame: Participants were tested twice with one week wash out (1h after having/skipping lunch)
Population: Complete case analysis
Measure: Median (Inter-Quartile Range); unit: Correct reactions
Arm/Group | Having Lunch | Skipping Lunch
Number analyzed (Participants) | 105 | 105
Correct reactions | 586 [533 to 656] | 594 [532 to 670]
Statistical Analysis 1: Comparison: Having Lunch vs Skipping Lunch; Test type: Non-Inferiority or Equivalence — No power calculation had been performed based on this measure; p = 0.45, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]

12. Primary Outcome: Incorrect Reactions
Description: Number of incorrect reactions
Time Frame: Participants were tested twice with one week wash out (1h after having/skipping lunch)
Population: Complete case analysis
Measure: Median (Inter-Quartile Range); unit: Incorrect reactions
Arm/Group | Having Lunch | Skipping Lunch
Number analyzed (Participants) | 105 | 105
Incorrect reactions | 30 [14 to 55] | 35 [19 to 59]
Statistical Analysis 1: Comparison: Having Lunch vs Skipping Lunch; Test type: Non-Inferiority or Equivalence — No power calculation had been performed based on this measure; p = 0.13, Wilcoxon (Mann-Whitney); [statistical method as in outcome 1, analysis 1]

13. Primary Outcome: Mean Time Correct Reactions
Description: Mean time to react correctly
Time Frame: Participants were tested twice with one week wash out (1h after having/skipping lunch)
Population: Complete case analysis
Measure: Median (Inter-Quartile Range); unit: Seconds
Arm/Group | Having Lunch | Skipping Lunch
Number analyzed (Participants) | 105 | 105
Seconds | 0.6 [0.6 to 0.7] | 0.6 [0.5 to 0.7]
Statistical Analysis 1: Comparison: Having Lunch vs Skipping Lunch; Test type: Non-Inferiority or Equivalence — No power calculation had been performed based on this measure; p = 0.68, Wilcoxon (Mann-Whitney); [statistical method as in outcome 1, analysis 1]

14. Primary Outcome: Mean Time Incorrect Reactions
Description: Mean time to react incorrectly
Time Frame: Participants were tested twice with one week wash out (1h after having/skipping lunch)
Population: Complete case analysis
Measure: Median (Inter-Quartile Range); unit: Seconds
Arm/Group | Having Lunch | Skipping Lunch
Number analyzed (Participants) | 105 | 105
Seconds | 0.5 [0.4 to 0.6] | 0.5 [0.4 to 0.6]
Statistical Analysis 1: Comparison: Having Lunch vs Skipping Lunch; Test type: Non-Inferiority or Equivalence — No power calculation had been performed based on this measure; p = 0.67, Wilcoxon (Mann-Whitney); [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Arm/Group | Having Lunch | Skipping Lunch
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/105
Other Adverse Events (participants affected / at risk) | 0/105 | 0/105

LIMITATIONS AND CAVEATS:
* Open-label study, in which everyone involved knew about group assignment
* Only one cognitive assessment per test day

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes